CLINICAL TRIAL: NCT06178991
Title: A PHASE 3, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A COMBINED MODIFIED RNA VACCINE CANDIDATE AGAINST COVID-19 AND INFLUENZA IN HEALTHY INDIVIDUALS
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Combined Modified RNA Vaccine Candidate Against COVID-19 and Influenza.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C5261002; NCT06178991 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-12-20; First posted 2023-12-21 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Influenza; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is an observer-blinded study. Study staff dispensing and administering the vaccine will be unblinded, but all other study personnel, including the principal investigator, and the participant, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 Arm A: Influenza and COVID-19 Combination A and Placebo (Experimental): Cohort 1 Arm A: Influenza and COVID-19 combination A vaccine and Placebo
  Interventions: Biological: Influenza and COVID-19 Combination A; Biological: Placebo
- Cohort 1 Arm B: COVID-19 vaccine and licensed influenza vaccine concomitant administration group (Active Comparator): Cohort 1 Arm B: COVID-19 vaccine and licensed influenza vaccine concomitant administration group
  Interventions: Biological: Licensed influenza vaccine; Biological: COVID-19 Vaccine
- Cohort 2 Arm C:Influenza and COVID-19 Combination B and Placebo (Experimental): Cohort 2 Arm C: Influenza and COVID-19 Combination B vaccine and Placebo
  Interventions: Biological: Influenza and COVID-19 Combination B; Biological: Placebo
- Cohort 2 Arm D: COVID-19 vaccine and licensed influenza vaccine concomitant administration group (Active Comparator): Cohort 2 Arm D: COVID-19 vaccine and licensed influenza vaccine concomitant administration group
  Interventions: Biological: Licensed influenza vaccine; Biological: COVID-19 Vaccine
- Cohort 3 Arm E:Influenza and COVID-19 Combination B (Experimental): Cohort 3 Arm E:Influenza and COVID-19 Combination B
  Interventions: Biological: Influenza and COVID-19 Combination B
- Cohort 3 Arm F: COVID-19 vaccine (Active Comparator): Cohort 3 Arm F: COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine
- Cohort 3 Arm G: Licensed influenza vaccine (Active Comparator): Cohort 3 Arm G: Licensed influenza vaccine
  Interventions: Biological: Licensed influenza vaccine
- Cohort 3 Arm H: Investigational influenza vaccine (Active Comparator): Cohort 3 Arm H: Investigational influenza vaccine
  Interventions: Biological: Investigational influenza vaccine

INTERVENTIONS:
Biological: Influenza and COVID-19 Combination A — Combined influenza and Pfizer-BioNTech COVID-19 Vaccine
  Arms: Cohort 1 Arm A: Influenza and COVID-19 Combination A and Placebo
Biological: Licensed influenza vaccine — Licensed influenza vaccine
  Arms: Cohort 1 Arm B: COVID-19 vaccine and licensed influenza vaccine concomitant administration group; Cohort 2 Arm D: COVID-19 vaccine and licensed influenza vaccine concomitant administration group; Cohort 3 Arm G: Licensed influenza vaccine
Biological: COVID-19 Vaccine — Pfizer-BioNTech COVID-19 vaccine
  Arms: Cohort 1 Arm B: COVID-19 vaccine and licensed influenza vaccine concomitant administration group; Cohort 2 Arm D: COVID-19 vaccine and licensed influenza vaccine concomitant administration group; Cohort 3 Arm F: COVID-19 vaccine
Biological: Influenza and COVID-19 Combination B — Combined influenza and Pfizer-BioNTech COVID-19 vaccine
  Arms: Cohort 2 Arm C:Influenza and COVID-19 Combination B and Placebo; Cohort 3 Arm E:Influenza and COVID-19 Combination B
Biological: Placebo — Saline Solution
  Arms: Cohort 1 Arm A: Influenza and COVID-19 Combination A and Placebo; Cohort 2 Arm C:Influenza and COVID-19 Combination B and Placebo
Biological: Investigational influenza vaccine — Investigational influenza vaccine
  Arms: Cohort 3 Arm H: Investigational influenza vaccine

SUMMARY:
The purpose of this study is to understand the safety and effects of a combined influenza and COVID-19 vaccine. This combined vaccine is compared to separate vaccines for the protection against influenza and SARS-CoV-2. Influenza and COVID-19 are diseases that can spread easily from one person to another and cause body aches, fever, cough, and other symptoms. Giving both influenza and COVID-19 vaccines together against influenza and SARS-CoV-2 could provide great benefits to both patients and caregivers in terms of simple and easy care. Around 8550 participants will be assigned into 1 of 8 vaccination groups (Group A, B, C, D, E, F, G or H) by chance.

Cohort 1: Approximately 450 participants will be assigned by chance to one of the following:

* Group A:Influenza and COVID-19 combination A vaccine, given at the same time in one arm and placebo (an injection consisting of just salt water and no medicines in it) in the opposite arm.
* Group B: COVID-19 vaccine, given at the same time to one arm and licensed influenza vaccine in the opposite arm.

Cohort 2: Approximately 4500 participants will be assigned by chance to one of the following:

* Group C: Influenza and COVID-19 combination B vaccine, given at the same time in one arm and placebo in the opposite arm.
* Group D: COVID-19 vaccine, given at the same time in one arm and licenced influenza vaccine in the opposite arm.

Cohort 3: Approximately 3600 participants will be assigned by chance to one of the following:

* Group E: Influenza and COVID-19 combination B vaccine.
* Group F: COVID-19 vaccine.
* Group G: Licenced influenza vaccine.
* Group H: Investigational influenza vaccine.

All participants in cohort 1 and cohort 2 will receive 2 injections and participants in cohort 3 will receive 1 injection as per their assigned study group at Visit 1. The participants will be followed for about 6 months. During this time, researchers will assess safety and the body's reaction to the vaccination over approximately 6 months. This will help understand if the study medicine is safe.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 through 64 years of age (or the minimum age of consent in accordance with local regulations) at Visit 1.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Exclusion Criteria:

* Vaccination with any investigational or licensed influenza vaccine within 6 months (175 days) before study intervention administration, or ongoing receipt of chronic antiviral therapy with activity against influenza.
* Vaccination with any investigational or licensed COVID-19 vaccine within 6 months (175 days) before study intervention administration.

Please refer to the study contact for further eligibility details

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8795 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (105):
- United States (105):
  - North Alabama Research Center, Athens, Alabama
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - AMR Clinical, Mobile, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Foothills Research Center/ CCT Research, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Baptist Health Center For Clinical Research, Little Rock, Arkansas
  - Hope Clinical Research, Inc., Canoga Park, California
  - Ascada Health PC dba Ascada Research, Fullerton, California
  - Orange County Research Center, Lake Forest, California
  - Ark Clinical Research, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Best Quality Research,Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Miami Clinical Research, Miami, Florida
  - Gerardo Polanco, MD, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Clinical Site Partners LLC, dba Flourish Research, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Angels Clinical Research Institute, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - AGILE Clinical Research Trials, LLC, Sandy Springs, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Prime, Idaho Falls, Idaho
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - AMR Clinical, Wichita, Kansas
  - Pharmaron, Baltimore, Maryland
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Headlands Research - Detroit, Southfield, Michigan
  - Revival Research Institute, LLC, Sterling Heights, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - McGill Family Practice, Papillion, Nebraska
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Rochester Clinical Research, LLC, Rochester, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare - Rocky Mount, Rocky Mount, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Mt. Auburn, Cincinnati, Ohio
  - Synexus Clinical Research US, Inc., Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Trial Management Associates, LLC, Myrtle Beach, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, Bristol, Tennessee
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research, LLC., Austin, Texas
  - Orion Clinical Research, Austin, Texas
  - Headlands Horizons, LLC dba Headlands Research-Brownsville, Brownsville, Texas
  - DFW Clinical Research, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Family Care, Fort Worth, Texas
  - Santa Clara Family Clinic, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - ACRC Trials (Administrative Location), Plano, Texas
  - ACRC TRIALS / North Texas Family Medicine, Plano, Texas
  - AIM Trials, LLC, Plano, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research, Martin Diagnostic Clinic, Tomball, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - AMR Clinical, Layton, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - AMR Clinical, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5261002

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo: Participants 18 to 64 years of age were administered with Influenza vaccine and coronavirus disease 2019 (COVID-19) vaccine (combination A) and placebo, intramuscularly on Day 1.
- Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration: Participants 18 to 64 years of age were administered concomitantly with COVID-19 vaccine and licensed influenza vaccine administered, intramuscularly on Day 1.
- Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo: Participants 18 to 64 years of age were administered with Influenza and COVID-19 vaccine (combination B) and placebo, intramuscularly on Day 1.
- Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B): Participants 18 to 64 years of age were administered with Influenza vaccine and COVID-19 vaccine (combination B), intramuscularly on Day 1.
- Cohort 3, Arm F: COVID-19 Vaccine: Participants 18 to 64 years of age were administered with COVID-19 vaccine, intramuscularly on Day 1.
- Cohort 3, Arm G: Licensed Influenza Vaccine: Participants 18 to 64 years of age were administered with licensed influenza vaccine, intramuscularly on Day 1.
- Cohort 3, Arm H: Investigational Influenza Vaccine: Participants 18 to 64 years of age were administered with investigational influenza vaccine, intramuscularly on Day 1.
Period: Overall Study
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Started (Randomized) | 313 | 160 | 3142 | 1572 | 1197 | 1195 | 607 | 609
Vaccinated | 309 | 159 | 3127 | 1563 | 1189 | 1191 | 605 | 607
Completed | 304 | 148 | 2938 | 1468 | 1110 | 1125 | 571 | 583
Not Completed | 9 | 12 | 204 | 104 | 87 | 70 | 36 | 26
Not completed — Withdrawal by Subject | 2 | 6 | 44 | 23 | 7 | 7 | 7 | 5
Not completed — Lost to Follow-up | 2 | 4 | 133 | 65 | 68 | 57 | 25 | 18
Not completed — Death | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Randomized but not Vaccinated | 4 | 1 | 15 | 9 | 8 | 4 | 2 | 2
Not completed — Other: Unspecified | 0 | 1 | 7 | 6 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was evaluated on safety population which included all participants who received at least 1 dose of the study intervention. Participants were grouped according to the vaccine as administered in the analysis based on the safety population.
Groups:
- Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo: Participants 18 to 64 years of age were administered with Influenza vaccine and COVID-19 vaccine (combination A) and placebo, intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine | Total
Number analyzed (Participants) | 309 | 159 | 3127 | 1563 | 1189 | 1191 | 605 | 607 | 8750
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (12.13) | 44.7 (13.89) | 44.0 (12.91) | 44.2 (12.53) | 44.3 (12.72) | 45.3 (12.45) | 44.5 (12.69) | 45.1 (12.82) | 44.4 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 95 | 1740 | 848 | 654 | 683 | 336 | 332 | 4868
  Male | 129 | 64 | 1387 | 715 | 535 | 508 | 269 | 275 | 3882
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 51 | 966 | 491 | 457 | 435 | 224 | 225 | 2954
  Not Hispanic or Latino | 201 | 108 | 2145 | 1055 | 719 | 739 | 372 | 371 | 5710
  Unknown or Not Reported | 3 | 0 | 16 | 17 | 13 | 17 | 9 | 11 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 22 | 17 | 13 | 4 | 4 | 2 | 63
  Asian | 4 | 6 | 111 | 58 | 35 | 34 | 18 | 20 | 286
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 12 | 2 | 9 | 3 | 2 | 2 | 31
  Black or African American | 74 | 37 | 812 | 392 | 277 | 295 | 143 | 157 | 2187
  White | 227 | 111 | 2106 | 1051 | 830 | 842 | 425 | 419 | 6011
  More than one race | 1 | 2 | 32 | 24 | 15 | 7 | 7 | 2 | 90
  Unknown or Not Reported | 2 | 2 | 32 | 19 | 10 | 6 | 6 | 5 | 82

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Percentage of Participants With Any Local Reactions for up to 7 Days Following Vaccination in Investigational Vaccine Extremity
Description: Local reactions included redness, swelling, and pain at the injection site, were recorded in the electronic dairy (e-diary) or case report form (CRF) after vaccination. Local reactions were graded per the 'Local Reaction Grading Scale' per protocol. Percentage of participants with at least 1 local reaction of grade 1 and above were reported in this outcome measure.
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day 1]
Population: Safety analysis population included all participants who received at least 1 dose of the study intervention. Participants were grouped according to the vaccine as administered in the analysis based on the safety population. Here "Overall Number of Participants Analyzed" signifies number of participants reporting at least 1 response in the e-diary or CRF after vaccination. As planned this outcome measure evaluated local reactions in investigational vaccine extremity.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 308 | 159
Percentage of participants | 74.7 [69.4 to 79.4] | 59.1 [51.1 to 66.8]

2. Primary Outcome: Cohort 2: Percentage of Participants With Any Local Reactions for up to 7 Days Following Vaccination in Investigational Vaccine Extremity
Description: Local reactions included redness, swelling, and pain at the injection site, were recorded in the e-diary or CRF after vaccination. Local reactions were graded per the 'Local Reaction Grading Scale' per protocol. Percentage of participants with at least 1 local reaction of grade 1 and above were reported in this outcome measure.
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day1]
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 3111 | 1560
Percentage of participants | 73.4 [71.8 to 75.0] | 63.5 [61.0 to 65.9]

3. Primary Outcome: Cohort 3: Percentage of Participants With Any Local Reactions for up to 7 Days Following Vaccination in Investigational Vaccine Extremity
Description: as for outcome 2
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day 1]
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Number analyzed (Participants) | 1186 | 1188 | 604 | 606
Percentage of participants | 73.4 [70.8 to 75.9] | 62.5 [59.6 to 65.2] | 34.8 [31.0 to 38.7] | 66.3 [62.4 to 70.1]

4. Primary Outcome: Cohort 1: Percentage of Participants With Any Systemic Events for up to 7 Days Following Vaccination
Description: Systemic events including fever, vomiting, diarrhea, headache, fatigue, chills, new or worsened muscle pain and new or worsened joint pain were recorded in an e-diary or CRF after vaccination. Systemic events were graded per the 'Systemic Events Grading Scale' per protocol. Percentage of participants with at least 1 systemic event of grade 1 and above were reported in this outcome measure.
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day 1]
Population: Safety analysis population included all participants who received at least 1 dose of the study intervention. Participants were grouped according to the vaccine as administered in the analysis based on the safety population. Here "Overall Number of Participants Analyzed" signifies number of participants reporting at least 1 response in the e-diary or CRF after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 308 | 159
Percentage of participants | 71.8 [66.4 to 76.7] | 54.1 [46.0 to 62.0]

5. Primary Outcome: Cohort 2: Percentage of Participants With Any Systemic Events for up to 7 Days Following Vaccination
Description: as for outcome 4
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day 1]
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 3111 | 1560
Percentage of participants | 70.8 [69.2 to 72.4] | 59.9 [57.4 to 62.3]

6. Primary Outcome: Cohort 3: Percentage of Participants With Any Systemic Events for up to 7 Days Following Vaccination
Description: as for outcome 4
Time Frame: From Day 1 through Day 7 after Vaccination [Vaccination on Day 1]
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Number analyzed (Participants) | 1186 | 1188 | 604 | 606
Percentage of participants | 66.7 [63.9 to 69.4] | 52.1 [49.2 to 55.0] | 43.9 [39.9 to 47.9] | 61.1 [57.0 to 65.0]

7. Primary Outcome: Cohort 1: Percentage of Participants Reporting Adverse Events (AEs) From Vaccination Through 4 Weeks After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious AEs. Serious AE (SAE) was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, any other pre-specified criteria in protocol of the study or other important medical event. Only AEs collected by non-systematic assessment (excluding local reactions and systematic events) were included in this outcome measure.
Time Frame: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: Safety analysis population included all participants who received at least 1 dose of the study intervention. Participants were grouped according to the vaccine as administered in the analysis based on the safety population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 309 | 159
Percentage of participants | 5.8 [3.5 to 9.1] | 10.1 [5.9 to 15.8]

8. Primary Outcome: Cohort 2: Percentage of Participants Reporting AEs From Vaccination Through 4 Weeks After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious AEs. SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, any other pre-specified criteria in protocol of the study or other important medical event. Only AEs collected by non-systematic assessment (excluding local reactions and systematic events) were included in this outcome measure.
Time Frame: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 3127 | 1563
Percentage of participants | 6.4 [5.6 to 7.3] | 6.1 [4.9 to 7.4]

9. Primary Outcome: Cohort 3: Percentage of Participants Reporting AEs From Vaccination Through 4 Weeks After Vaccination
Description: as for outcome 8
Time Frame: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Number analyzed (Participants) | 1189 | 1191 | 605 | 607
Percentage of participants | 3.8 [2.8 to 5.0] | 4.8 [3.6 to 6.2] | 4.1 [2.7 to 6.0] | 4.1 [2.7 to 6.0]

10. Primary Outcome: Cohort 1: Percentage of Participants Reporting SAEs From Vaccination Through 6 Months After Vaccination
Description: SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, and any other pre-specified criteria in protocol of the study or other important medical event.
Time Frame: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 309 | 159
Percentage of participants | 0.6 [0.1 to 2.3] | 2.5 [0.7 to 6.3]

11. Primary Outcome: Cohort 2: Percentage of Participants Reporting SAEs From Vaccination Through 6 Months After Vaccination
Description: as for outcome 10
Time Frame: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 3127 | 1563
Percentage of participants | 0.7 [0.5 to 1.1] | 1.4 [0.9 to 2.1]

12. Primary Outcome: Cohort 3: Percentage of Participants Reporting SAEs From Vaccination Through 6 Months After Vaccination
Description: as for outcome 10
Time Frame: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Number analyzed (Participants) | 1189 | 1191 | 605 | 607
Percentage of participants | 0.8 [0.4 to 1.5] | 1.3 [0.7 to 2.1] | 0.8 [0.3 to 1.9] | 1.2 [0.5 to 2.4]

13. Primary Outcome: Cohort 2: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Strain-Specific Hemagglutination Inhibition Assay (HAI) Titers at 4 Weeks After Vaccination: Non-inferiority
Description: GMTs and the corresponding 2-sided confidence interval (CIs) were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the lower limit of quantitation (LLOQ) were set to 0.5 *LLOQ. GMTs were reported in the descriptive data section of this outcome measure. GMRs were reported in the statistical analysis section. Data was reported for the following strains: H1N1, H3N2 and Victoria.
Time Frame: At 4 Weeks after Vaccination
Population: Evaluable immunogenicity population (EIP): eligible participants, received study intervention per randomization, had minimum 1 valid and determinate immunogenicity result from blood sample collected within 27- 42 days postvaccination, and had no major protocol violations. EIP for HAI of Cohort 2 was utilized. "Number Analyzed": participants evaluable for specific strains. All participants for "Overall Number of Participants Analyzed" added to the data but may not be present as "Number Analyzed".
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 1923 | 967
Titer
  H1N1: number analyzed (Participants) | 1916 | 964
  H1N1 | 188.3 [178.2 to 198.9] | 136.3 [125.9 to 147.5]
  H3N2: number analyzed (Participants) | 1909 | 954
  H3N2 | 165.9 [158.0 to 174.1] | 96.9 [90.6 to 103.5]
  Victoria: number analyzed (Participants) | 1918 | 965
  Victoria | 37.4 [35.5 to 39.5] | 56.4 [52.4 to 60.6]
Statistical Analysis 1: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; H1N1; Test type: Non-Inferiority — The criterion for non-inferiority (NI) was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.38, 95% CI 2-sided [1.25 to 1.52] — GMRs (ratio of Arm C to Arm D titers) and 2-sided 95% CIs were calculated by exponentiating mean difference of the logarithms of the titers between the two comparative vaccine groups and the corresponding CIs (based on the Student t distribution)
Statistical Analysis 2: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; H3N2; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.71, 95% CI 2-sided [1.58 to 1.86] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; Victoria; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 0.66, 95% CI 2-sided [0.61 to 0.73] — [estimate comment as in outcome 13, analysis 1]

14. Primary Outcome: Cohort 2: Percentage of Participants and Difference in Percentage of Participants With Strain-Specific HAI Seroconversion at 4 Weeks After Vaccination: Non-inferiority
Description: Seroconversion was defined as having an HAI titer <1:10 prior to vaccination and greater than or equal to (>=) 1:40 at the postvaccination time point of interest, or an HAI titer of >=1:10 prior to vaccination with a minimum 4-fold rise at the postvaccination time point of interest. Percentage of participants with seroconversion were reported in the descriptive data section of this outcome measure. Difference in percentage of participants with seroconversion were reported in the statistical analysis section. Data was reported for the following strains: H1N1, H3N2 and Victoria.
Time Frame: At 4 Weeks after Vaccination
Population: EIP: eligible participants, received study intervention per randomization, had minimum 1 valid and determinate immunogenicity result from blood sample collected within 27- 42 days postvaccination, and had no major protocol violations. EIP for HAI of Cohort 2 was utilized. "Number Analyzed": participants evaluable for specific strains. All participants for "Overall Number of Participants Analyzed" added to the data but may not be present as "Number Analyzed".
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 1923 | 967
Percentage of participants
  H1N1: number analyzed (Participants) | 1913 | 958
  H1N1 | 72.8 [70.7 to 74.8] | 54.9 [51.7 to 58.1]
  H3N2: number analyzed (Participants) | 1887 | 943
  H3N2 | 65.7 [63.5 to 67.8] | 40.1 [36.9 to 43.3]
  Victoria: number analyzed (Participants) | 1915 | 962
  Victoria | 31.7 [29.6 to 33.8] | 45.4 [42.2 to 48.6]
Statistical Analysis 1: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; H1N1; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the difference in percentage of participants achieving seroconversion was greater than -10%; Difference in percentage of participants = 17.9, 95% CI 2-sided [14.1 to 21.6] — Difference in percentage of participants achieving seroconversion (Arm C - Arm D) and the associated 2-sided 95% CI was based on the Miettinen and Nurminen method. Data was expressed as percentages
Statistical Analysis 2: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; H3N2; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Difference in percentage of participants = 25.6, 95% CI 2-sided [21.7 to 29.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; Victoria; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Difference in percentage of participants = -13.7, 95% CI 2-sided [-17.5 to -10.0] — [estimate comment as in outcome 14, analysis 1]

15. Primary Outcome: Cohort 2: GMT and GMR of Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Neutralizing Titers at 4 Weeks After Vaccination: Non-inferiority
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5 *LLOQ. GMTs were reported in the descriptive data section of this outcome measure. GMRs were reported in the statistical analysis section.
Time Frame: At 4 Weeks after Vaccination
Population: EIP: eligible participants, received study intervention per randomization, had minimum 1 valid and determinate immunogenicity result from blood sample collected within 27- 42 days postvaccination, and had no major protocol violations. EIP for SARS-CoV-2 neutralization of Cohort 2 was utilized. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 2941 | 1480
Titer | 3535.1 [3370.0 to 3708.4] | 3476.6 [3256.7 to 3711.4]
Statistical Analysis 1: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.02, 95% CI 2-sided [0.94 to 1.10] — [estimate comment as in outcome 13, analysis 1]

16. Primary Outcome: Cohort 2: Percentage of Participants and Difference in Percentage of Participants With SARS-CoV-2 Seroresponse at 4 Weeks After Vaccination: Non-inferiority
Description: Seroresponse was defined as achieving a postvaccination >=4-fold rise from baseline (before the study vaccination). If the baseline measurement was below the LLOQ, the postvaccination measure of >=4*LLOQ was considered seroresponse. Percentage of participants with seroresponse were reported in the descriptive data section of this outcome measure. Difference in percentage of participants with seroresponse were reported in the statistical analysis section.
Time Frame: At 4 Weeks after Vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration
Number analyzed (Participants) | 2932 | 1473
Percentage of participants | 75.5 [73.9 to 77.1] | 73.7 [71.4 to 76.0]
Statistical Analysis 1: Comparison: Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo vs Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the difference in percentage of participants achieving seroresponse was greater than -10%; Difference in percentage of participants = 1.8, 95% CI 2-sided [-0.9 to 4.6] — Difference in percentage of participants achieving seroresponse (Arm C - Arm D) and the associated 2-sided 95% CI was based on the Miettinen and Nurminen method. Data was expressed as percentages

17. Secondary Outcome: Cohort 3: GMT and GMR of Strain-Specific HAI Titers at 4 Weeks After Vaccination: Non-inferiority
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5 *LLOQ. GMTs were reported in the descriptive data section of this outcome measure. GMRs were reported in the statistical analysis section. Data was reported for reported for following strains: H1N1, H3N2 and Victoria.
Time Frame: At 4 Weeks after Vaccination
Population: EIP:eligible participants, received study intervention per randomization, had minimum 1 valid and determinate immunogenicity result from blood sample collected within 27- 42 days postvaccination, and had no major protocol violations. EIP for HAI of Cohort 3 was utilized. "Overall Number of Participants Analyzed": participants evaluable for this outcome; "Number Analyzed": participants evaluable at specific strains. Per plan only those arms where influenza vaccine was administered were evaluated.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
Number analyzed (Participants) | 1132 | 579 | 580
Titer
  H1N1: number analyzed (Participants) | 1132 | 577 | 580
  H1N1 | 165.6 [153.5 to 178.7] | 142.5 [126.9 to 160.0] | 170.2 [153.2 to 189.2]
  H3N2: number analyzed (Participants) | 1124 | 572 | 580
  H3N2 | 175.7 [165.3 to 186.8] | 100.1 [90.9 to 110.3] | 190.4 [173.4 to 209.2]
  Victoria | 39.2 [36.6 to 42.1] | 67.4 [61.1 to 74.3] | 31.5 [28.6 to 34.6]
Statistical Analysis 1: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm G: Licensed Influenza Vaccine; H1N1; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.16, 95% CI 2-sided [1.01 to 1.34] — GMRs (ratio of Arm E to Arm G titers) and 2-sided 95% CIs were calculated by exponentiating mean difference of the logarithms of the titers between the two comparative vaccine groups and the corresponding CIs (based on the Student t distribution)
Statistical Analysis 2: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm H: Investigational Influenza Vaccine; H1N1; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 0.97, 95% CI 2-sided [0.85 to 1.11] — GMRs (ratio of Arm E to Arm H titers) and 2-sided 95% CIs were calculated by exponentiating mean difference of the logarithms of the titers between the two comparative vaccine groups and the corresponding CIs (based on the Student t distribution)
Statistical Analysis 3: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm G: Licensed Influenza Vaccine; H3N2; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.75, 95% CI 2-sided [1.56 to 1.97] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm H: Investigational Influenza Vaccine; H3N2; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 0.92, 95% CI 2-sided [0.82 to 1.03] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 5: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm G: Licensed Influenza Vaccine; Victoria; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 0.58, 95% CI 2-sided [0.52 to 0.66] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm H: Investigational Influenza Vaccine; Victoria; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 1.25, 95% CI 2-sided [1.11 to 1.40] — [estimate comment as in outcome 17, analysis 2]

18. Secondary Outcome: Cohort 3: GMT and GMR of SARS-CoV-2 Neutralizing Titers at 4 Weeks After Vaccination: Non-inferiority
Description: as for outcome 15
Time Frame: At 4 Weeks after Vaccination
Population: EIP: eligible participants, received study intervention per randomization, had minimum 1 valid and determinate immunogenicity result from blood sample collected within 27-42 days postvaccination, and had no major protocol violations. EIP for SARS-CoV-2 neutralization of Cohort 3 was utilized. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure. Per plan only those arms where COVID-19 vaccine was administered were evaluated.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine
Number analyzed (Participants) | 1120 | 1135
Titer | 3841.0 [3577.3 to 4124.1] | 4208.9 [3901.8 to 4540.2]
Statistical Analysis 1: Comparison: Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) vs Cohort 3, Arm F: COVID-19 Vaccine; Test type: Non-Inferiority — The criterion for NI was lower bounds of the 2-sided 95% CI for the GMR was greater than 0.67; GMR = 0.91, 95% CI 2-sided [0.82 to 1.01] — GMRs (ratio of Arm E to Arm F titers) and 2-sided 95% CIs were calculated by exponentiating mean difference of the logarithms of the titers between the two comparative vaccine groups and the corresponding CIs (based on the Student t distribution)

ADVERSE EVENTS:
Time Frame: Systematic assessment: Local reactions and systemic events were assessed from Vaccination on Day 1 to Day 7 after Vaccination; Non-systematic assessment: all-cause mortality and SAEs were assessed from Vaccination on Day 1 up to 6 months after Vaccination; other AEs were assessed from Vaccination on Day 1 up to 4 weeks after Vaccination
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis population included all participants who received at least 1 dose of the study intervention.
Arm/Group | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) | Cohort 3, Arm F: COVID-19 Vaccine | Cohort 3, Arm G: Licensed Influenza Vaccine | Cohort 3, Arm H: Investigational Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 1/309 | 0/159 | 2/3127 | 1/1563 | 1/1189 | 0/1191 | 1/605 | 1/607
Serious Adverse Events (participants affected / at risk) | 2/309 | 4/159 | 23/3127 | 22/1563 | 10/1189 | 15/1191 | 5/605 | 7/607
Other Adverse Events (participants affected / at risk) | 245/309 | 113/159 | 2521/3127 | 1152/1563 | 941/1189 | 843/1191 | 330/605 | 456/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo (N=309) | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration (N=159) | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo (N=3127) | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration (N=1563) | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) (N=1189) | Cohort 3, Arm F: COVID-19 Vaccine (N=1191) | Cohort 3, Arm G: Licensed Influenza Vaccine (N=605) | Cohort 3, Arm H: Investigational Influenza Vaccine (N=607)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute cardiac event (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Device related bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Arm A: Influenza Vaccine and COVID-19 Vaccine (Combination A) and Placebo (N=309) | Cohort 1, Arm B: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration (N=159) | Cohort 2, Arm C: Influenza Vaccine and COVID-19 Vaccine (Combination B) and Placebo (N=3127) | Cohort 2, Arm D: COVID-19 Vaccine and Licensed Influenza Vaccine Concomitant Administration (N=1563) | Cohort 3, Arm E: Influenza Vaccine and COVID-19 Vaccine (Combination B) (N=1189) | Cohort 3, Arm F: COVID-19 Vaccine (N=1191) | Cohort 3, Arm G: Licensed Influenza Vaccine (N=605) | Cohort 3, Arm H: Investigational Influenza Vaccine (N=607)
COVID-19 (Infections and infestations) | 1 | 2 | 15 | 10 | 2 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 15 | 17 | 3 | 6 | 1 | 3
Chills (CHILLS) (General disorders) | 117 | 26 | 1163 | 295 | 327 | 144 | 40 | 133
Fatigue (FATIGUE) (General disorders) | 180 | 66 | 1780 | 705 | 610 | 448 | 186 | 289
Injection site erythema (REDNESS) (General disorders) | 44 | 11 | 293 | 103 | 122 | 84 | 18 | 46
Injection site pain (PAIN) (General disorders) | 227 | 93 | 2259 | 976 | 861 | 732 | 199 | 396
Injection site swelling (SWELLING) (General disorders) | 40 | 12 | 376 | 122 | 151 | 101 | 20 | 62
Pyrexia (FEVER) (General disorders) | 43 | 4 | 331 | 71 | 123 | 30 | 6 | 35
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 45 | 22 | 446 | 207 | 164 | 140 | 64 | 77
Vomiting (VOMITING) (Gastrointestinal disorders) | 12 | 3 | 123 | 48 | 51 | 30 | 12 | 12
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 77 | 18 | 640 | 212 | 220 | 128 | 45 | 94
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 114 | 23 | 1081 | 368 | 356 | 214 | 62 | 167
Headache (HEADACHE) (Nervous system disorders) | 147 | 47 | 1403 | 517 | 489 | 343 | 145 | 197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (or its agents) has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT06178991/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT06178991/SAP_001.pdf